CLINICAL TRIAL: NCT03969940
Title: Thermotherapy of Buruli Ulcer at Community Level in the Health District of Akonolinga
Acronym: UB Thermo
Status: Withdrawn | Type: Observational
Why Stopped: Lack of supply of comparator drug in country
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: University Hospital Heidelberg (Other); Centre International de Recherches, d'Enseignements et de Soins (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2018-13
Record Dates: First submitted 2019-05-23; First posted 2019-05-31 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-11

CONDITIONS: Buruli Ulcer
MeSH Terms: conditions — Buruli Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thermo: Buruli ulcer patients receiving thermotherapy
- Chemo: Buruli ulcer patients receiving chemotherapy

SUMMARY:
The project rolls out combined innovative low-tech thermotherapy of Buruli ulcer (BU) with heat packs and WHO recommended wound management in a BU endemic district of Cameroon.

DETAILED DESCRIPTION:
The project translates available clinical research findings at the secondary health care level into clinical practice at the primary health care and community level. The string of previous work from the development of the BU thermotherapy-wound management-package to the proof of its efficacy provides all necessary procedures, tools and documents to immediately proceed into practical and integrated community application.

Main objective:

To determine in patients with early BU lesions the effectiveness and acceptability of thermotherapy treatment at health post and community level.

Specific objectives:

1. To monitor and evaluate clinical and biological responses to thermotherapy in patients receiving up to 8 weeks of thermotherapy
2. To assess within 6 months after completion of heat treatment wound closure ("primary cure") and/or absence of BU specific features in included patients according to WHO healing criteria
3. To measure the BU recurrence rate in included patient within 12 months after completion of heat treatment' ("definite cure").
4. To assess the compliance rate of included patients
5. To assess the withdrawal rate of included patients
6. To assess the ability and comfort of health personnel to use the thermotherapy device

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed BU patients with a single WHO category I and II lesion

Exclusion Criteria:

- inappropriate lesion size (category III patients), location and patients with multiple lesions

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include inhabitants of all health areas of the Akonolinga health district or coming from other BU endemic areas of Cameroon.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary cure: wound closure and/or no BU features according to WHO guideline | 6 months
  Number of patients with wound closure and/or absence of clinically BU specific features according to WHO guidelines within 6 months after completion of heat treatment
Definite cure: No recurrence | 12 months
  Number of patients with no BU recurrence for 12 months after completion of heat treatment

SECONDARY OUTCOMES:
Acceptability | 2 years
  Rates of withdrawal (due to low compliance or consent withdrawal)
Acceptability | 2 years
  Rating of thermotherapy by health staff

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Junghanss, MD, Study Chair — University Hospital Heidelberg

IPD SHARING:
Plan to Share IPD: No